CLINICAL TRIAL: NCT03401853
Title: Phase II Study of Anti-CD20 Antibody Therapy Plus Pembrolizumab (MK-3475) in Subjects With Relapsed Follicular and Diffuse Large B-Cell Lymphoma
Brief Title: Pembrolizumab With Rituximab or Obinutuzumab in Treating Patients With Relapsed or Refractory Follicular Lymphoma or Diffuse Large B Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated to end of funding.
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Stephen Smith, Associate Professor, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9469; NCI-2017-02361 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9469 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1717070 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma
Keywords: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — pembrolizumab; Rituximab; CT-P10; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (pembrolizumab, rituximab) (Experimental): INDUCTION: Patients diagnosed with R/R FL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Biological: Rituximab
- Arm II (pembrolizumab, rituximab) (Experimental): INDUCTION: Patients diagnosed with R/R DLBCL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Biological: Rituximab
- Arm III (pembrolizumab, obinutuzumab) (Experimental): INDUCTION: Patients diagnosed with R/R FL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive obinutuzumab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Biological: Obinutuzumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83; rituximab biosimilar TQB2303; rituximab-abbs; Truxima; Rituximab Biosimilar SIBP-02
  Arms: Arm I (pembrolizumab, rituximab); Arm II (pembrolizumab, rituximab)
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759
  Arms: Arm III (pembrolizumab, obinutuzumab)

SUMMARY:
This phase II trial studies how well pembrolizumab with rituximab or obinutuzumab work in treating patients with follicular lymphoma or diffuse large B cell lymphoma that has come back (recurrent) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Rituximab and obinutuzumab are monoclonal antibodies. They bind to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Giving pembrolizumab with rituximab or obinutuzumab may help kill more cancer cells in patients with follicular lymphoma or diffuse large B cell lymphoma.

DETAILED DESCRIPTION:
OUTLINE: Patients are assigned to 1 of 3 arms.

ARM I:

INDUCTION: Patients diagnosed with R/R FL receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.

EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.

ARM II:

INDUCTION: Patients diagnosed with R/R DLBCL receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.

EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.

Arm III:

INDUCTION: Patients diagnosed with R/R FL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive obinutuzumab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.

EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity. Patients with stable disease or better, who are experiencing clinical benefit in the judgment of the investigator, may receive obinutuzumab IV on day 1 of cycles 5, 9, 13, 17, 21, and 25.

After completion of study treatment, patients are followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Have relapsed/refractory DLBCL or relapsed/refractory FL

  * For DLBCL, patients must have relapsed after, declined, or considered ineligible for high-dose chemotherapy and autologous stem cell transplantation
  * For FL, in addition to relapsed/refractory disease status, patients must have received therapy with CD20 antibody-directed therapy, and must have an indication for treatment; FL eligibility also requires patients have no standard options with curative potential, nor options with more favorable risk/benefit ratio in the judgment of the investigator
  * For FL Arm C (obinutuzumab + pembrolizumab), patients must have relapsed/refractory disease after rituximab-containing therapy including:

    * Rituximab in combination with chemotherapy (at 1 prior line) or
    * >= 2 prior lines of therapy
    * Patients may have no standard options with curative potential, nor options with more favorable risk/benefit ratio in the judgment of the investigator
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease (1.5 cm or greater in the longest diameter of nodal or extranodal disease)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 500/uL (within 28 days of cycle 1 day 1)

  * Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed
  * No lower limit if cytopenia is related to bone marrow involvement
* Platelets >= 25,000/uL (within 28 days of cycle 1 day 1)

  * Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed
  * No lower limit if cytopenia is related to bone marrow involvement
* Hemoglobin >= 8 g/dL (within 28 days of cycle 1 day 1)

  * Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed
  * No lower limit if cytopenia is related to bone marrow involvement
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for subject with creatinine levels > 1.5 X institutional ULN (within 28 days of cycle 1 day 1)

  **Creatinine clearance (CrCl) should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 X ULN (within 28 days of cycle 1 day 1)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver involvement by lymphoma (within 28 days of cycle 1 day 1)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 28 days of cycle 1 day 1)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 28 days of cycle 1 day 1)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception; contraception, for the course of the study until at least 12 months after the last dose of study medication

  **Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy until at least 12 months after the last dose of study therapy

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment, except for physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency which is permitted
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Prior allogeneic transplant, within the last 5 years
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study

  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or lymphomatous meningitis; subjects with previously treated brain metastases or lymphomatous meningitis may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through until at least 12 months after the last dose of study treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy. Administration of killed vaccines is allowed

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Smith, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I Follicular Lymphoma (Pembrolizumab, Rituximab): INDUCTION: Patients diagnosed with R/R FL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Rituximab: Given IV
- Arm II DLBCL (Pembrolizumab, Rituximab): INDUCTION: Patients diagnosed with R/R DLBCL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Rituximab: Given IV
- Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab): INDUCTION: Patients diagnosed with R/R FL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive obinutuzumab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity. Patients with stable disease or better, who are experiencing clinical benefit in the judgment of the investigator, may receive obinutuzumab IV on day 1 of cycles 5, 9, 13, 17, 21, and 25.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Obinutuzumab: Given IV
Period: Overall Study
Arm/Group | Arm I Follicular Lymphoma (Pembrolizumab, Rituximab) | Arm II DLBCL (Pembrolizumab, Rituximab) | Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab)
Started | 7 | 8 | 3
Completed | 7 | 8 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm II DLBCL (Pembrolizumab, Obinutuzumab): INDUCTION: Patients diagnosed with R/R DLBCL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Rituximab: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm I Follicular Lymphoma (Pembrolizumab, Rituximab) | Arm II DLBCL (Pembrolizumab, Obinutuzumab) | Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab) | Total
Number analyzed (Participants) | 7 | 8 | 3 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 2 | 9
  >=65 years | 1 | 7 | 1 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 5
  Male | 4 | 6 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 6 | 8 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 8 | 3 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Will be defined as the rate of complete + partial responses using computed tomography (CT) criteria (Lugano 2014).
Time Frame: Up to 90 days after the last dose of pembrolizumab
Measure: Number; unit: percentage of participants
Groups:
- Arm I Follicular Lymphoma (Pembrolizumab, Rituximab): INDUCTION: Patients with R/R FL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Rituximab: Given IV
- Arm II DLBCL (Pembrolizumab, Rituximab): INDUCTION: Patients with R/R DLBCL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Rituximab: Given IV
- Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab): INDUCTION: Patients with R/R FL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive obinutuzumab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity. Patients with stable disease or better, who are experiencing clinical benefit in the judgment of the investigator, may receive obinutuzumab IV on day 1 of cycles 5, 9, 13, 17, 21, and 25.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Obinutuzumab: Given IV
Arm/Group | Arm I Follicular Lymphoma (Pembrolizumab, Rituximab) | Arm II DLBCL (Pembrolizumab, Rituximab) | Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab)
Number analyzed (Participants) | 7 | 8 | 3
percentage of participants | 29 | 0 | 0

2. Secondary Outcome: Incidence of Serious or Drug-related Adverse Events
Description: Evaluated by the NCI Common Terminology for Adverse Events (CTCAE), version 4.0.
Time Frame: Up to 90 days after the last dose of pembrolizumab
Measure: Number; unit: percentage of participants
Arm/Group | Arm I Follicular Lymphoma (Pembrolizumab, Rituximab) | Arm II DLBCL (Pembrolizumab, Rituximab) | Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab)
Number analyzed (Participants) | 7 | 8 | 3
percentage of participants | 100 | 63 | 67

3. Secondary Outcome: Progression-free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate median PFS.
Time Frame: Up to 90 days after the last dose of pembrolizumab
Measure: Median (80% Confidence Interval); unit: years
Groups:
- Arm II DLBCL (Pembrolizumab, Obinutuzumab): INDUCTION: Patients with R/R DLBCL receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, and 15 of cycle 1, and on day 1 of cycle 2.
  EXTENDED THERAPY: Patients with at least a partial response receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (35 cycles) in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Rituximab: Given IV
Arm/Group | Arm I Follicular Lymphoma (Pembrolizumab, Rituximab) | Arm II DLBCL (Pembrolizumab, Obinutuzumab) | Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab)
Number analyzed (Participants) | 7 | 8 | 3
years | 0.23 [0.18 to NA] — Upper bound could not be calculated due to insufficient number of participants with events. | 0.21 [0.11 to NA] — Upper bound could not be calculated due to insufficient number of participants with events.. | 0.50 [0.38 to NA] — Upper bound could not be calculated due to insufficient number of participants with events..

4. Secondary Outcome: Overall Survival (OS)
Description: The Kaplan-Meier method will be used to estimate median OS.
Time Frame: Up to 90 days after the last dose of pembrolizumab
Measure: Median (80% Confidence Interval); unit: years
Arm/Group | Arm I Follicular Lymphoma (Pembrolizumab, Rituximab) | Arm II DLBCL (Pembrolizumab, Obinutuzumab) | Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab)
Number analyzed (Participants) | 7 | 8 | 3
years | NA [3.1 to NA] — Median and upper bound could not be calculated due to insufficient number of participants with events.. | 1.5 [0.65 to NA] — Upper bound could not be calculated due to insufficient number of participants with events.. | NA [1.1 to NA] — Median and upper bound could not be calculated due to insufficient number of participants with events..

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of informed consent and for 90 days after the last dose of pembrolizumab.
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Arm/Group | Arm I Follicular Lymphoma (Pembrolizumab, Rituximab) | Arm II DLBCL (Pembrolizumab, Rituximab) | Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab)
All-Cause Mortality (participants affected / at risk) | 2/7 | 5/8 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/7 | 5/8 | 0/3
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Follicular Lymphoma (Pembrolizumab, Rituximab) (N=7) | Arm II DLBCL (Pembrolizumab, Rituximab) (N=8) | Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab) (N=3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Altered mental status (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Streptococcus salivarius (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Follicular Lymphoma (Pembrolizumab, Rituximab) (N=7) | Arm II DLBCL (Pembrolizumab, Rituximab) (N=8) | Arm III Follicular Lymphoma (Pembrolizumab, Obinutuzumab) (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (4) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Creatinine Increased (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Fatigue (Gastrointestinal disorders) | 5 (5) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Infusion related reaction (General disorders) | 3 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lower extremity pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Attention deficit hyperactive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin - Hands (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythematous rash, flanks (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
small white bumps on lips (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Alopecia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Edema Limbs (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Right leg swelling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized Tingling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot Flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Investigations) | 0 (0) | 1 (1) | 0 (0)
muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Right Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus, Adenovirus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Foot Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03401853/Prot_SAP_001.pdf